CLINICAL TRIAL: NCT01473888
Title: An Open-label, One-sequence, Two Periods, Crossover Trial Study to Evaluate the Effect of T89 on the Pharmacokinetics of Five CYP450 Substrates Cocktail in Healthy Subjects
Brief Title: A Study To Evaluate The Effect of T89(Dantonic®)On P450 Enzymes
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Tasly Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None
Other Study IDs: T89-02-US
Record Dates: First submitted 2011-10-31; First posted 2011-11-17 (Estimated); Last update posted 2012-11-08 (Estimated); Status verified 2011-11

CONDITIONS: Stable Angina
Keywords: T89(Dantonic®); Cooperstown 5+1 cocktail probes; CYP450
MeSH Terms: conditions — Angina, Stable | interventions — T89 herbal drug

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- T89 (Other)
  Interventions: Drug: T89(Dantonic)

INTERVENTIONS:
Drug: T89(Dantonic) — capsule, 225mg B.I.D.

SUMMARY:
Purpose: This study is to determine the effect of T89(Dantonic®)on P450 enzymes. This study will help determine which types of drugs may interact with T89.

DETAILED DESCRIPTION:
T89 is a modernized and industrialized version of a traditional Chinese herbal medicine. T89 was approved for marketing as a drug, for the treatment of chronic stable angina pectoris due to coronary heart disease, by the State Food and Drug Administration (SFDA) of China in 1993. There were more than 2 billion doses have been prescribed or used, in about 10,000,000 subjects, in short or long-term administration worldwide.

The product is also marketed, as a drug, in Russia, South Korea, Mongolia, Singapore, Vietnam, and South Africa. The current study is to determine the anti-angina effect and dose response of T89 in patients with chronic stable angina pectoris in the United States.

T89 consists of Danshen (Radix Salviae Miltiorrhizae, RSM) and Sanqi (Radix Notoginseng, RN) as active constitutes, and using Borneol as transporting enhancer.

ELIGIBILITY:
Inclusion Criteria:

* Nonsmoking Male or female 18-50 years of age, with a body mass index (BMI)18 to ≤ 30 kg/m2
* Healthy adult with no active medical problems or significant chronic diseases as determined by the study doctor based on history, physical exam and laboratory evaluations;
* Avoid eating Seville oranges, grapefruits (including grapefruit juice), broccoli, brussels sprouts, charcoal-grilled meats, alcoholic beverages, and caffeine- and theobromine-containing beverages and foods for the duration of the study beginning at the screening visit.
* Females of child bearing potential must be able to maintain adequate birth control during the study; defined as double barrier method or complete abstinence. Females of non-child bearing potential must provide documentation of tubal ligation or hysterectomy.
* Be able to provide written informed consent and comply with requirements of the study;
* Be able to read, speak and understand English

Exclusion Criteria:

* Clinically significant abnormal findings by history, physical exam, ECG, or laboratory testing as determined by the study doctor.
* Know hypersensitivity or intolerance to any of the probe substrates or the active and/or inactive ingredients in the probe substrates, flumazenil, guaifenesin, or vitamin K;
* A history of illicit drug use or a history of alcohol abuse within 1 year of screening.
* Women who are pregnant, breastfeeding, and/or not using an acceptable form of non-hormonal contraception (double barrier method or abstinence) during the study.
* History of gastrointestinal bleeding or peptic ulcer disease.
* Any condition that may affect drug absorption (e.g., gastrectomy, malabsorption syndromes).
* Had an elevated international normalized ratio (INR) time (INR> 1.2) at screening or Day-1.
* Had taken any nicotine-containing or nicotine replacement devices within 6 months before the screening visit
* Had taken any prescription drugs during the 3 months before the screening visit
* Had taken any nonprescription drugs (including natural health products, Vitamins, and herbals) during a period of 7 days prior to the screening visit
* Had received an immunization during the 2 weeks prior to the screening visit
* Had known immune deficiency disease or were positive for human immunodeficiency virus, Hepatitis B or Hepatitis C virus.
* Use of any drug known to inhibit or induce hepatic enzymes within 30 days of the first study phase.
* Regular alcohol intake exceeding 1 drink/day (1 drink = 5 ounces of wine or 12 ounces of beer or 1 ounce of hard liquor) within 7 days of screening.
* Treatment with an investigational drug within 30 days or 5 half-lives (whichever is longer) preceding the first dose of study drug.
* Presence of any condition that the investigator feels would interfere with successful completion of the study.
* Genotyping of poor metabolizers for CYP2D6, CYP2C9, and CYP2C19.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2011-01; Primary Completion 2011-07 (Actual); Study Completion 2012-01 (Actual)

PRIMARY OUTCOMES:
The PK variables of the cocktail substrates with and without T89. | 25 days (From Day 1 to Day 25)
  caffine: AUC(0-12h)&Cmax; Omeprazole:AUC(0-12h)& Cmax; Midazolam:AUC(0-12h)& Cmax; Dextromethorphan:Dextromethorphan/Dextrorphan(12h Urine)
  S-warfarin: AUC(0-96h)& Cmax;

SECONDARY OUTCOMES:
Safety assessments (AEs, Vital signs, ECG, Safety labs, INRs) | subjects will be followed for the safety assessment from Day 0 to Day 35.

CONTACTS AND LOCATIONS:
Overall Officials: Jason Zhixin GUO, M.D., Study Director — Tasly Pharmaceuticals Co. Ltd.
Locations (1):
- Comprehensive Clinical Development NW Inc., Tacoma, Washington, United States

REFERENCES:
- See also: Related Info — http://www.tasly.com